CLINICAL TRIAL: NCT01958788
Title: Challenging Uncertainty: Behavioural Experiments in the Treatment of Generalized Anxiety Disorder
Brief Title: Testing Beliefs About Uncertainty in the Treatment of Generalized Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Concordia University, Montreal (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Principal Investigator, Elizabeth A. Hebert, M.A., Ph.D. Candidate, Concordia University, Montreal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOP-69066-620
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Results first posted 2016-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-01

CONDITIONS: Generalized Anxiety Disorder
Keywords: Cognitive-behavioral treatment; Generalized anxiety disorder; Worry; Behavioral experiments; Safety behaviors; Anxiety
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cognitive-Behavioural Treatment (Experimental): 12 sessions of cognitive-behavioral treatment targeting negative beliefs about uncertainty
  Interventions: Behavioral: Cognitive-Behavioural Treatment

INTERVENTIONS:
Behavioral: Cognitive-Behavioural Treatment — 12 weekly sessions of individual cognitive-behavioural treatment (CBT) targeting intolerance of uncertainty.

SUMMARY:
Generalized Anxiety Disorder (GAD) is an anxiety disorder characterized by excessive and uncontrollable worry. Our research group has developed a cognitive-behavioural treatment (CBT) for GAD centered upon intolerance of uncertainty, a dispositional characteristic that arises from a set of negative beliefs about uncertainty and its consequences (Dugas & Robichaud, 2007). This CBT protocol has demonstrated good efficacy over four previous clinical trials: approximately 70% of participants fully remit from GAD following treatment and maintain these gains over extended follow-up periods. These results, while positive, do suggest that a substantial minority of individuals do not fully benefit from the existing treatment protocol. Across our randomized clinical trials, individuals who do not achieve diagnostic remission of GAD continue to endorse elevated levels of intolerance of uncertainty. This suggests that the current CBT protocol does not effectively reduce intolerance of uncertainty in some treated individuals. To address this, we have developed a modified version of the original CBT protocol that targets intolerance of uncertainty more directly. The goal of the current proposal is to determine whether this newly developed CBT protocol with fewer components can deliver comparable or superior GAD symptom reduction. A total of 7 participants with a primary diagnosis of GAD received the newly developed CBT protocol over 12 weekly sessions. Measures of GAD symptoms, psychopathology, and intolerance of uncertainty were administered at pre-, mid-, and post-treatment, as well as at 3- and 6-month follow-ups. The proposed study will provide information about the efficacy of this new CBT protocol in reducing GAD symptoms.

DETAILED DESCRIPTION:
Generalized anxiety disorder (GAD) is characterized by excessive and uncontrollable worry and anxiety. This common and debilitating anxiety disorder is associated with significant distress as well as substantial impairment in occupational, social, and daily functioning. As a result, effective treatment for GAD is essential. Several cognitive-behavioural treatment (CBT) protocols have been developed for GAD, including an efficacious treatment developed by our research group. This CBT protocol for GAD centres upon intolerance of uncertainty, a dispositional characteristic that arises from a set of negative beliefs about uncertainty and its consequences (Dugas & Robichaud, 2007). Previous research has shown that individuals with GAD demonstrate high intolerance of uncertainty, and that there are a number of potential pathways by which intolerance of uncertainty may lead to symptoms of GAD (see Dugas & Robichaud, 2007 for a review). Our CBT protocol targeting intolerance of uncertainty has demonstrated good efficacy across four published randomized clinical trials: approximately 70% of participants have fully remitted from GAD following treatment and have maintained these gains over extended follow-up periods. These results, while positive, do suggest that a substantial minority of individuals do not fully benefit from the existing treatment protocol. Across our randomized clinical trials, individuals who do not achieve diagnostic remission of GAD continue to endorse elevated levels of intolerance of uncertainty. This suggests that the current CBT protocol does not effectively reduce intolerance of uncertainty in some treated individuals. Additionally, the existing treatment protocol has 6 major components, utilizes a number of cognitive and behavioural techniques (including symptom monitoring, motivational interviewing, situational exposure, problem-solving training, and imaginal exposure), and requires at least 14 sessions to implement. Recent literature (e.g., Cougle et al., 2011) has suggested that there is increased need for parsimony and efficiency in CBT protocols. As a result, our research group is investigating new methods of targeting intolerance of uncertainty that demonstrate greater parsimony and efficiency.

Our previous CBT protocol for GAD targeted intolerance of uncertainty directly through situational exposure, and indirectly through motivational interviewing, problem-solving training, and imaginal exposure. In an effort to streamline and strengthen GAD treatment, the newly developed CBT protocol only targets intolerance of uncertainty directly. In this new CBT protocol, intolerance of uncertainty was targeted using behavioural experiments in which participants identified and tested out their beliefs about uncertainty. The extant literature suggests that behavioural experiments are an efficacious way to target the emotional, cognitive, and behavioural components of anxiety disorders and may be superior to habituation-based exposure paradigms (McMillan & Lee, 2010; Salkovskis et al., 2007).

The current study examined if a newly developed CBT protocol with fewer components could deliver comparable GAD symptom reduction. Seven (7) individuals with a primary diagnosis of GAD completed 12 sessions of CBT using a newly developed treatment protocol focusing exclusively on intolerance of uncertainty. The treatment consisted of 50-minute, weekly sessions targeting intolerance of uncertainty primarily via behavioural experiments. The three treatment components included: (1) psychoeducation and uncertainty awareness training; (2) testing beliefs about uncertainty (via behavioural experiments); and (3) relapse prevention. Measures of GAD symptoms, general psychopathology, and intolerance of uncertainty were administered at pre-, mid-, and post-treatment, as well as at 3- and 6-month follow-ups. Our main outcomes of interest were effect sizes (i.e., relative magnitude of change from pre-posttreatment, pretreatment to 6-month follow-up, and posttreatment to 6-month follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of GAD (as assessed by semi-structured clinical interviews)
* Score of 58 or greater on the (Intolerance of Uncertainty Scale)
* Willingness to keep medication status stable while participating in the study

Exclusion Criteria:

* Change in medication type or dose in 12 weeks before study entry
* Use of herbal products known to have central nervous system effects in the 2 weeks before study entry
* Evidence of suicidal intent
* Evidence of current substance abuse
* Evidence of current or past schizophrenia, bipolar disorder or organic mental disorder
* Current participation in other trials
* Concurrent psychotherapy during treatment phase of trial
* Evidence of anxiety symptoms due to a general medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Hebert, M.A., Principal Investigator — Concordia University, Montreal
Locations (1):
- Concordia University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was approved by Human Research Ethics Committees of Concordia University and the Hôpital du Sacré-Coeur de Montréal. Participants self-referred to the Hôpital du Sacré-Coeur de Montréal anxiety clinic via advertisements placed in a local newspaper. Recruitment occurred between April 2013 to March 2014.
Groups:
- Cognitive-Behavioural Treatment: 12 weekly sessions of individual cognitive-behavioural treatment (CBT) targeting intolerance of uncertainty via behavioural experiments.
Period: Overall Study
Arm/Group | Cognitive-Behavioural Treatment
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cognitive-Behavioural Treatment
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 7

OUTCOME MEASURES:

1. Primary Outcome: Clinician's Severity Rating (CSR) Scale of Anxiety Disorders Interview Schedule for DSM-IV (ADIS-IV)
Description: The CSR is a severity rating scale ranging from 0-8. Scores of 4 or greater represent clinically significant symptoms, whereas scores lower than 4 indicate subclinical symptoms. Lower scores represent improved outcome. This measure was used to evaluate change from baseline in the severity of GAD symptoms as assessed by the ADIS-IV, a semi-structured clinical interview for Axis I disorders.
Time Frame: Pretreatment to posttreatment (12 weeks) and 6-month Follow-Up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive-Behavioural Treatment
Number analyzed (Participants) | 7
units on a scale
  Pretreatment ADIS-IV | 5.5 (0.82)
  Posttreatment ADIS-IV | 3.14 (1.03)
  6-month follow-up ADIS-IV | 2.43 (1.90)
Statistical Analysis 1: Comparison: Cognitive-Behavioural Treatment; Pre-posttreatment effect size estimation using Cohen's d: a calculation of the relative magnitude of the effect from pretreatment to posttreatment; Test type: Superiority or Other; Cohen's d effect size; Cohen's d effect size = 2.06
Statistical Analysis 2: Comparison: Cognitive-Behavioural Treatment; Pretreatment to 6-month follow-up effect size estimation using Cohen's d: a calculation of the relative magnitude of the effect from pretreatment to 6-month follow-up; Test type: Superiority or Other; Cohen's d effect size; Cohen's d effect size = 1.34
Statistical Analysis 3: Comparison: Cognitive-Behavioural Treatment; Posttreatment to 6-month follow-up effect size estimation using Cohen's d: a calculation of the relative magnitude of the effect from posttreatment to 6-month follow-up; Test type: Superiority or Other; Cohen's d effect size; Cohen's d effect size = 0.37

2. Secondary Outcome: Worry and Anxiety Questionnaire (WAQ)
Description: The WAQ is a questionnaire assessing self-reported symptoms of GAD. Scores range from 0 to 56, with higher scores indicating greater severity of self-rated GAD symptoms. The measure was used to assess change from baseline in self-reported GAD symptoms (WAQ).
Time Frame: Pretreatment to posttreatment (12 weeks) and 6-month Follow-Up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive-Behavioural Treatment
Number analyzed (Participants) | 7
units on a scale
  Pretreatment WAQ | 38.36 (5.25)
  Posttreatment WAQ | 24.36 (9.06)
  6-month follow-up WAQ | 25.43 (6.42)
Statistical Analysis 1: Comparison: Cognitive-Behavioural Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Cohen's d effect size; Cohen's d effect size = 1.32
Statistical Analysis 2: Comparison: Cognitive-Behavioural Treatment; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Cohen's d effect size; Cohen's d effect size = 1.29
Statistical Analysis 3: Comparison: Cognitive-Behavioural Treatment; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; Cohen's d effect size; Cohen's d effect size = -0.15

3. Secondary Outcome: Intolerance of Uncertainty Scale (IUS)
Description: The IUS is a self-report questionnaire assessing intolerance of uncertainty, or the tendency to view uncertainty and its consequences as negative. Scores range from 27 to 135, with higher scores representing greater intolerance of uncertainty. The IUS was used to assess change from baseline in self-reported intolerance of uncertainty.
Time Frame: Pretreatment to posttreatment (12 weeks) and 6-month Follow-Up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive-Behavioural Treatment
Number analyzed (Participants) | 7
units on a scale
  Pretreatment IUS | 85.71 (14.71)
  Posttreatment IUS | 55.00 (15.55)
  6-month follow-up IUS | 54.29 (12.30)
Statistical Analysis 1: Comparison: Cognitive-Behavioural Treatment; Pre-posttreatment follow-up effect size estimation using Cohen's d: a calculation of the relative magnitude of the effect from pretreatment to posttreatment follow-up; Test type: Superiority or Other; Cohen's d effect size; Cohen's d effect size = 1.72
Statistical Analysis 2: Comparison: Cognitive-Behavioural Treatment; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Cohen's d effect size; Cohen's d effect size = 1.66
Statistical Analysis 3: Comparison: Cognitive-Behavioural Treatment; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; Cohen's d effect size; Cohen's d effect size = 0.07

4. Secondary Outcome: Penn State Worry Questionnaire (PSWQ)
Description: The PSWQ is a self-report questionnaire assessing excessive and uncontrollable worry. Scores range from 16 to 80, with greater scores indicating greater worry. The PSWQ was used to evaluate change from baseline in self-reported worry.
Time Frame: Pretreatment to posttreatment (12 weeks) and 6-month Follow-Up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive-Behavioural Treatment
Number analyzed (Participants) | 7
units on a scale
  Pretreatment PSWQ | 61.57 (6.00)
  Posttreatment PSWQ | 50.00 (8.25)
  6-month follow-up PSWQ | 51.14 (6.15)
Statistical Analysis 1: Comparison: Cognitive-Behavioural Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Cohen's d effect size; Cohen's d effect size = 1.13
Statistical Analysis 2: Comparison: Cognitive-Behavioural Treatment; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Cohen's d effect size; Cohen's d effect size = 1.06
Statistical Analysis 3: Comparison: Cognitive-Behavioural Treatment; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; Cohen's d effect size; Cohen's d effect size = -0.18

5. Secondary Outcome: GAD Safety Behaviours Questionnaire (GAD-SBQ)
Description: The GAD-SBQ is a self-report questionnaire assessing the tendency to use safety behaviours to cope with anxiety, such as reassurance-seeking and overpreparation. Scores range from 18 to 90, with greater scores indicating greater use of safety behaviours. The GA-SBQ was used to evaluate change from baseline in self-reported safety behaviours.
Time Frame: Pretreatment to posttreatment (12 weeks) and 6-month Follow-Up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive-Behavioural Treatment
Number analyzed (Participants) | 7
units on a scale
  Pretreatment GAD-SBQ | 47.00 (9.95)
  Posttreatment GAD-SBQ | 32.71 (5.53)
  6-month follow-up GAD-SBQ | 36.14 (5.11)
Statistical Analysis 1: Comparison: Cognitive-Behavioural Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Cohen's d effect size; Cohen's d effect size = 1.41
Statistical Analysis 2: Comparison: Cognitive-Behavioural Treatment; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Cohen's d effect size; Cohen's d effect size = 1.65
Statistical Analysis 3: Comparison: Cognitive-Behavioural Treatment; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; Cohen's d effect size; Cohen's d effect size = -0.70

6. Secondary Outcome: Beck Anxiety Inventory (BAI)
Description: The BAI is a self-report questionnaire assessing affective, cognitive, and somatic anxiety over the preceding week. Scores range from 0 to 63, with greater scores representing greater self-reported anxiety. The BAI was used to evaluate change from baseline in self-reported anxiety.
Time Frame: Pretreatment to posttreatment (12 weeks) and 6-month Follow-Up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive-Behavioural Treatment
Number analyzed (Participants) | 7
units on a scale
  Pretreatment BAI | 23.71 (10.47)
  Posttreatment BAI | 9.86 (10.56)
  6-month follow-up BAI | 12.57 (12.12)
Statistical Analysis 1: Comparison: Cognitive-Behavioural Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Cohen's d effect size; Cohen's d effect size = 1.64
Statistical Analysis 2: Comparison: Cognitive-Behavioural Treatment; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Cohen's d effect size; Cohen's d effect size = 1.47
Statistical Analysis 3: Comparison: Cognitive-Behavioural Treatment; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; Cohen's d effect size; Cohen's d effect size = -0.56

7. Secondary Outcome: Beck Depression Inventory, 2nd Edition (BDI-II)
Description: The BDI-II is a self-report questionnaire assessing a variety of depressive symptoms, including low mood, anhedonia, and worthlessness. Scores range from 0 to 63, with greater scores indicating greater depressive symptoms. The BDI-II was used to evaluate change from baseline in self-reported depressive symptoms.
Time Frame: Pretreatment to posttreatment (12 weeks) and 6-month Follow-Up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive-Behavioural Treatment
Number analyzed (Participants) | 7
units on a scale
  Pretreatment BDI-II | 14.71 (4.39)
  Posttreatment BDI-II | 4.00 (5.69)
  6-month follow-up BDI-II | 5.57 (5.16)
Statistical Analysis 1: Comparison: Cognitive-Behavioural Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Cohen's d effect size; Cohen's d effect size = 2.08
Statistical Analysis 2: Comparison: Cognitive-Behavioural Treatment; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Cohen's d effect size; Cohen's d effect size = 2.15
Statistical Analysis 3: Comparison: Cognitive-Behavioural Treatment; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; Cohen's d effect size; Cohen's d effect size = -0.55

ADVERSE EVENTS:
Time Frame: 9 months per participant (12 weeks treatment, 6-month follow-up)
Description: Participant's mental health status was assessed at pretreatment, midtreatment, posttreatment, 3-month follow-up, and 6-month follow-up.
Arm/Group | Cognitive-Behavioural Treatment
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
Small sample size due to clinical case replication series design. This reduced statistical power and types of statistical analyses that could be conducted. Participants were homogeneous in ethnicity and language, which may limit generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No